CLINICAL TRIAL: NCT00004848
Title: A Controlled Prospective Study of Transfusion-Associated Hepatitis
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 810110; 81-CC-0110
Record Dates: First submitted 2000-03-02; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-07

CONDITIONS: Hepatitis
Keywords: AIDS; Autologous Blood; Cardiac Surgery; HIV; Hepatocellular Inflammation; Liver Biopsy; Long Term Sera Storage; Non-A Hepatitis; Non-B Hepatitis
MeSH Terms: conditions — Hepatitis; Acquired Immunodeficiency Syndrome; Hepatitis C

SUMMARY:
This protocol represents a continuation of a series of prospective studies to define the incidence and etiology of transfusion-associated hepatitis (TAH) and to examine the impact on TAH of various modifications in the selection of blood donors.

The primary goal of the study will be to determine TAH incidence after the institution of a variety of interventive measures to exclude hepatitis and AIDS virus carriers: including surrogate assays (ALT, anti-HBc), a specific assay for the hepatitis C virus (HCV), a specific assay for the human immunodeficiency virus (HIV) and intensified donor questioning for high-risk behavior patterns. There is high probability that the exclusion of donors at high risk for AIDS transmission will also exclude donors at high risk for hepatitis transmission.

Incidence data obtained in the study will be enhanced by the simultaneous follow-up of a control population undergoing identical surgical procedures, but receiving no blood or only autologous blood. This control population, made possible by the recent dramatic increase in the amount of autologous blood utilized, will allow for a clear distinction between transfusion-associated hepatitis and that due to nosocomial transmission or other background causes of hepatocellular inflammation in cardiac surgery patients.

DETAILED DESCRIPTION:
This protocol represents a continuation of a series of prospective studies to define the incidence and etiology of transfusion-associated hepatitis (TAH) and to examine the impact on TAH of various modifications in the selection of blood donors.

The primary goal of the study will be to determine TAH incidence after the institution of a variety of interventive measures to exclude hepatitis and AIDS virus carriers: including surrogate assays (ALT, anti-HBc), a specific assay for the hepatitis C virus (HCV), a specific assay for the human immunodeficiency virus (HIV) and intensified donor questioning for high-risk behavior patterns. There is high probability that the exclusion of donors at high risk for AIDS transmission will also exclude donors at high risk for hepatitis transmission.

Incidence data obtained in the study will be enhanced by the simultaneous follow-up of a control population undergoing identical surgical procedures, but receiving no blood or only autologous blood. This control population, made possible by the recent dramatic increase in the amount of autologous blood utilized, will allow for a clear distinction between transfusion-associated hepatitis and that due to nosocomial transmission or other background causes of hepatocellular inflammation in cardiac surgery patients.

ELIGIBILITY:
Consecutive patients undergoing open-heart surgery at Georgetown University and Fairfax Hospital will be admitted to the study if:

They are 18 years of age or older;

They provide informed consent;

They reside in the United States and will be available for at least six months of follow up.

Patients with known hepatitis C or hepatitis B virus carriers with or without evidence of chronic hepatitis will be excluded.

Persons with a history of prior hepatitis will not be excluded, but will be analyzed as a separate cohort.

Patients with close exposure (household or sexual contact) to hepatitis in the preceding six months will be excluded.

Patients with elevated pre-operative alanine aminotransferase (ALT) will be excluded. An aspartate aminotransferase (AST) of between 45 and 75 IU per L will not serve as cause for exclusion if the corresponding ALT is normal on at least two occasions.

A preoperative AST greater than 75 IU/L will serve to exclude patients from study independent of the ALT.

Patients with blood transfusion in the six months preceding surgery will be excluded. Patients will also be retrospectively excluded if they receive blood more than one month after surgery.

The six month followup period will be timed from the date of the last transfusion.

Patients with alcoholism or other known liver or active biliary tract disease at the time of entrance into the study will be excluded.

Patients with inadequate veins from which to obtain required samples will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 1981-07; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Stevens CE, Aach RD, Hollinger FB, Mosley JW, Szmuness W, Kahn R, Werch J, Edwards V. Hepatitis B virus antibody in blood donors and the occurrence of non-A, non-B hepatitis in transfusion recipients. An analysis of the Transfusion-Transmitted Viruses Study. Ann Intern Med. 1984 Dec;101(6):733-8. doi: 10.7326/0003-4819-101-6-733. PMID 6437308
- [Background] Koziol DE, Holland PV, Alling DW, Melpolder JC, Solomon RE, Purcell RH, Hudson LM, Shoup FJ, Krakauer H, Alter HJ. Antibody to hepatitis B core antigen as a paradoxical marker for non-A, non-B hepatitis agents in donated blood. Ann Intern Med. 1986 Apr;104(4):488-95. doi: 10.7326/0003-4819-104-4-488. PMID 3006567